CLINICAL TRIAL: NCT01771627
Title: Pilot Study of Varenicline vs. Nicotine Patch Delivered by a Telephone Quitline to Promote Smoking Cessation
Brief Title: Varenicline or Nicotine Patch in Promoting Smoking Cessation Among Current Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I 221312; NCI-2012-02755 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Results first posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Varenicline; Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (varenicline) (Experimental): Patients undergo general smoking cessation counseling and receive varenicline PO QD on days 1-28. Courses repeat every 28 days for up to 12 weeks.
  Interventions: Drug: varenicline
- Arm II (nicotine patch) (Active Comparator): Patients undergo general smoking cessation counseling and receive nicotine patch continuously for 12 weeks.
  Interventions: Drug: nicotine patch

INTERVENTIONS:
Drug: varenicline — Given PO
  Other Names: Champix; Chantix; CP-526555
  Arms: Arm I (varenicline)
Drug: nicotine patch
  Other Names: NicoDerm CQ; nicotine skin patch; nicotine transdermal patch; nicotine transdermal system patch
  Arms: Arm II (nicotine patch)

SUMMARY:
This pilot clinical trial studies varenicline or nicotine patch in promoting smoking cessation among current smokers. Varenicline or nicotine patch may help people stop smoking

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if mail delivery of 12 weeks of varenicline results in improved smoking cessation outcomes relative to nicotine replacement therapy (NRT) in 300 smokers.

II. To determine if delivery of varenicline is cost-effective as compared to nicotine patch.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo general smoking cessation counseling and receive varenicline orally (PO) twice daily (QD) on days 1-28. Courses repeat every 28 days for up to 12 weeks.

ARM II: Patients undergo general smoking cessation counseling and receive nicotine patch continuously for 12 weeks.

After completion of study treatment, patients are followed up at 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Cigarette smokers who call the New York State Smokers' Quitline requesting assistance with quitting smoking
* State that they are under the care of a primary care physician
* Are eligible for receipt of pharmacotherapy by mail using the standard NRT criteria
* Speak English
* Answer "no" to the following 3 questions:

  * "Have you ever been diagnosed with or treated for a mental health problem like major depression, bipolar disorder, dysthymia, or schizoaffective disorder?"
  * "Have you ever had serious thoughts of killing or hurting yourself, ever have any intention or plan to carry out these thoughts, or actually attempted to kill yourself?"
  * "Is there any reason that you cannot use varenicline/Chantix?"

Exclusion Criteria:

* State that they are not under the care of a primary care physician
* Are not eligible for receipt of pharmacotherapy by mail using the standard NRT criteria
* Do not speak English
* Answer "yes" to the question, "have you ever been diagnosed with or treated for a mental health problem like major depression, bipolar disorder, dysthymia, or schizoaffective disorder?"
* Answer "yes" to the question, "have you ever had serious thoughts of killing or hurting yourself, ever have any intention or plan to carry out these thoughts, or actually attempted to kill yourself?"
* Answer "yes" to the question, "is there any reason that you cannot use varenicline/Chantix?"
* Are women who are currently pregnant
* Report that they are unwilling to receive or take varenicline on screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-10-22 (Actual); Primary Completion 2014-09-28 (Actual); Study Completion 2015-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Mahoney, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
available upon request from PI
Supporting Information: Study Protocol
Time Frame: now thru 2021
Access Criteria: available upon request from PI

REFERENCES:
- [Background] Rojewski AM, Hyland A, Mahoney MC. Cooper LM, Zuromski KL, Celestino P, Koutsky J, Toll BA. Feasibility of delivering varenicline through a telephone quitline to promote smoking cessation. J Smoking Cessation 2018
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm II (Nicotine Patch): Patients undergo general smoking cessation counseling and receive nicotine patch continuously for 12 weeks.
  nicotine patch
Period: Overall Study
Arm/Group | Arm I (Varenicline) | Arm II (Nicotine Patch)
Started | 200 | 100
Completed | 92 | 50
Not Completed | 108 | 50

BASELINE CHARACTERISTICS:
Population: VAR: mean age 47, 77% white, 10% Hispanic, 46% female NRT: mean age 46, 84% white, 13% Hispanic, 47% female
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Varenicline) | Arm II (Nicotine Patch) | Total
Number analyzed (Participants) | 200 | 100 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 200 | 100 | 300
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (13.9) | 46.1 (13.8) | 47 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 47 | 140
  Male | 107 | 53 | 160
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 13 | 34
  Not Hispanic or Latino | 179 | 87 | 266
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 46 | 16 | 62
  White | 154 | 84 | 238
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 200 | 100 | 300

OUTCOME MEASURES:

1. Primary Outcome: Quit Rate
Description: The quit rate at 4 months will be compared between the 2 groups, using a logistic regression analysis with a 2-side 95% confidence interval.
Time Frame: 4 months
Population: self reported abstinence
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Varenicline) | Arm II (Nicotine Patch)
Number analyzed (Participants) | 36 | 50
Participants | 13 | 23

ADVERSE EVENTS:
Arm/Group | Arm I (Varenicline) | Arm II (Nicotine Patch)
All-Cause Mortality (participants affected / at risk) | 0/200 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/200 | 0/100
Other Adverse Events (participants affected / at risk) | 0/200 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes